CLINICAL TRIAL: NCT02294474
Title: Six-month, Randomized, Open-label, Parallel-group Comparison of the Insulin Analog SAR342434 to Humalog® in Adult Patients With Type 2 Diabetes Mellitus Also Using Insulin Glargine
Brief Title: Comparison of SAR342434 to Humalog as the Rapid Acting Insulin in Adult Patients With Type 2 Diabetes Mellitus Also Using Insulin Glargine
Acronym: SORELLA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC13403; 2014-002844-42 (EudraCT Number); U1111-1156-4296 (UTN)
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SAR342434; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR342434 (Experimental): SAR342434 100 Unit/mL (U/mL) before meals intake on top of once daily (QD) Insulin Glargine, up to Week 26.
  Interventions: Drug: SAR342434; Drug: insulin glargine HOE901
- Humalog (Active Comparator): Humalog 100 U/mL before meals intake on top of QD Insulin Glargine, up to Week 26.
  Interventions: Drug: Humalog; Drug: insulin glargine HOE901

INTERVENTIONS:
Drug: SAR342434 — SAR342434 100 U/mL (dose range of 1 Unit to 80 Units) self-administered by subcutaneous (SC) injection, immediately (within 5 -10 minutes) before meals intake. Dose adjusted to achieve 2 hour post prandial glucose (PPG) in range of 6.7 to 8.9 mmol/L (120 to 160 mg/dL) while avoiding hypoglycemia.
  Arms: SAR342434
Drug: Humalog — Humalog 100 U/ml (dose range of 1 unit to 60 units) self-administered by SC injection, immediately (within 5-10 minutes) before meals intake. Dose adjusted to achieve a 2 hour PPG in range of 6.7 to 8.9 mmol/L (120 to 160 mg/dL) while avoiding hypoglycemia.
  Other Names: Insulin Lispro
  Arms: Humalog
Drug: insulin glargine HOE901 — Insulin glargine 100 U/mL injected QD subcutaneously consistent with the local label. Doses adjusted to achieve glycemic target for fasting, preprandial plasma glucose (SMPG) between 4.4 to 7.2 mmol/L (80 to 130 mg/dL) without hypoglycemia.
  Other Names: Lantus®

SUMMARY:
Primary Objective:

To demonstrate non-inferiority of SAR342434 versus Humalog in glycated hemoglobin A1c (HbA1c) change from baseline to Week 26 in participants with type 2 diabetes mellitus (T2DM) also using insulin glargine.

Secondary Objectives:

To assess the immunogenicity of SAR342434 and Humalog in terms of positive/negative status and antibody titers at baseline and during the course of the study; To assess the relationship of anti-insulin antibodies with efficacy and safety. To assess the efficacy of SAR342434 and Humalog on: proportion of participants reaching target HbA1c <7.0% and <=6.5%, fasting plasma glucose (FPG) and self-measured plasma glucose (SMPG) profiles, and insulin dose.

To assess safety of SAR342434 and Humalog.

DETAILED DESCRIPTION:
The study will consist of a: up to 2 weeks screening period, 26-week treatment period, and 1-day follow-up period.

The maximum study duration will then be 28 weeks per participant and a 1-day safety follow-up.

ELIGIBILITY:
Inclusion criteria:

* Participants with T2DM diagnosed for at least 12 months and treated with insulin glargine and Humalog®/Liprolog® or NovoLog®/NovoRapid® (at least 3 times daily, before each meal) in the 6 months prior to the screening visit.
* Signed written informed consent.

Exclusion criteria:

* At screening visit, age under legal age of adulthood.
* HbA1c <6.5% or >10.0% at screening.
* Diabetes other than T2DM.
* Pregnancy and lactation.
* Women of childbearing potential not protected by highly effective contraceptive method of birth control.
* Use of insulin pump in the 6 months before screening visit.
* Use of insulin other than insulin glargine and Humalog or NovoLog/NovoRapid in the 6 months prior to screening visit. Liprolog® is an European Union (EU) approved insulin lispro and is allowed in those countries where it is marketed.
* Use of Humalog/Liprolog or Novolog/NovoRapid less than 3 times daily, before each meal.
* Use of non-injectable peptides (eg, Glucagon-like peptide-1 (GLP-1) receptor-agonists or other peptides) in the 6 months prior to screening visit.
* Body mass index (BMI) >=40kg/m² at screening visit.
* Hospitalization for diabetic ketoacidosis in the last 6 months before screening visit.
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment, or injectable drugs) during the study period.
* The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (103):
- United States (51):
  - Investigational Site Number 840217, Foley, Alabama
  - Investigational Site Number 840237, Muscle Shoals, Alabama
  - Investigational Site Number 840245, Chandler, Arizona
  - Investigational Site Number 840219, Phoenix, Arizona
  - Investigational Site Number 840227, Phoenix, Arizona
  - Investigational Site Number 840212, Little Rock, Arkansas
  - Investigational Site Number 840241, El Cajon, California
  - Investigational Site Number 840238, Fresno, California
  - Investigational Site Number 840229, Greenbrae, California
  - Investigational Site Number 840231, Huntington Beach, California
  - Investigational Site Number 840247, Long Beach, California
  - Investigational Site Number 840234, Los Angeles, California
  - Investigational Site Number 840235, Northridge, California
  - Investigational Site Number 840251, Palm Springs, California
  - Investigational Site Number 840249, Santa Ana, California
  - Investigational Site Number 840223, Temecula, California
  - Investigational Site Number 840259, Tustin, California
  - Investigational Site Number 840240, Walnut Creek, California
  - Investigational Site Number 840214, Boynton Beach, Florida
  - Investigational Site Number 840246, Miami, Florida
  - Investigational Site Number 840226, New Port Richey, Florida
  - Investigational Site Number 840205, Ocoee, Florida
  - Investigational Site Number 840206, Palm Harbor, Florida
  - Investigational Site Number 840242, Port Charlotte, Florida
  - Investigational Site Number 840253, Lawrenceville, Georgia
  - Investigational Site Number 840207, Stockbridge, Georgia
  - Investigational Site Number 840248, Arlington Heights, Illinois
  - Investigational Site Number 840204, Avon, Indiana
  - Investigational Site Number 840257, Evansville, Indiana
  - Investigational Site Number 840230, Des Moines, Iowa
  - Investigational Site Number 840239, Rockville, Maryland
  - Investigational Site Number 840236, Troy, Michigan
  - Investigational Site Number 840216, Lincoln, Nebraska
  - Investigational Site Number 840220, Las Vegas, Nevada
  - Investigational Site Number 840233, Las Vegas, Nevada
  - Investigational Site Number 840224, Linden, New Jersey
  - Investigational Site Number 840232, Greensboro, North Carolina
  - Investigational Site Number 840211, Morehead City, North Carolina
  - Investigational Site Number 840228, Morganton, North Carolina
  - Investigational Site Number 840225, Fargo, North Dakota
  - Investigational Site Number 840221, Columbus, Ohio
  - Investigational Site Number 840255, Dayton, Ohio
  - Investigational Site Number 840250, Tipton, Pennsylvania
  - Investigational Site Number 840243, Uniontown, Pennsylvania
  - Investigational Site Number 840208, Chattanooga, Tennessee
  - Investigational Site Number 840215, Jackson, Tennessee
  - Investigational Site Number 840203, Austin, Texas
  - Investigational Site Number 840258, Dallas, Texas
  - Investigational Site Number 840201, Dallas, Texas
  - Investigational Site Number 840222, Renton, Washington
  - Investigational Site Number 840209, Milwaukee, Wisconsin
- Argentina (5):
  - Investigational Site Number 032201, Caba
  - Investigational Site Number 032206, Capital Federal
  - Investigational Site Number 032202, Capital Federal
  - Investigational Site Number 032205, Ciudad Autonoma de Buenos Aire
  - Investigational Site Number 032203, Salta
- Chile (3):
  - Investigational Site Number 152202, Santiago
  - Investigational Site Number 152204, Santiago
  - Investigational Site Number 152201, Santiago
- Investigational Site Number 170203, Armenia, Colombia
- Germany (6):
  - Investigational Site Number 276201, Berlin
  - Investigational Site Number 276204, Heidelberg
  - Investigational Site Number 276202, Neumünster
  - Investigational Site Number 276206, Potsdam
  - Investigational Site Number 276205, Stuttgart
  - Investigational Site Number 276203, Sulzbach-Rosenberg
- Hungary (7):
  - Investigational Site Number 348205, Budapest
  - Investigational Site Number 348202, Budapest
  - Investigational Site Number 348204, Debrecen
  - Investigational Site Number 348208, Komárom
  - Investigational Site Number 348210, Nagykanizsa
  - Investigational Site Number 348209, Sátoraljaújhely
  - Investigational Site Number 348203, Szolnok
- Italy (4):
  - Investigational Site Number 380203, Bologna
  - Investigational Site Number 380201, Milan
  - Investigational Site Number 380204, Roma
  - Investigational Site Number 380202, Sesto San Giovanni
- Romania (10):
  - Investigational Site Number 642210, Bacau
  - Investigational Site Number 642201, Bucharest
  - Investigational Site Number 642202, Bucharest
  - Investigational Site Number 642206, Cluj-Napoca
  - Investigational Site Number 642204, Deva
  - Investigational Site Number 642205, Oradea
  - Investigational Site Number 642209, Sibiu
  - Investigational Site Number 642207, Târgu Mureş
  - Investigational Site Number 642208, Târgu Mureş
  - Investigational Site Number 642203, Timișoara
- Russia (5):
  - Investigational Site Number 643201, Saint Petersburg
  - Investigational Site Number 643203, Saint Petersburg
  - Investigational Site Number 643204, Saint Petersburg
  - Investigational Site Number 643202, Saint Petersburg
  - Investigational Site Number 643205, Saratov
- South Korea (4):
  - Investigational Site Number 410202, Seoul
  - Investigational Site Number 410204, Seoul
  - Investigational Site Number 410205, Seoul
  - Investigational Site Number 410201, Wŏnju
- Spain (3):
  - Investigational Site Number 724201, Barcelona
  - Investigational Site Number 724203, Málaga
  - Investigational Site Number 724202, Palma de Mallorca
- Turkey (Türkiye) (4):
  - Investigational Site Number 792201, Istanbul
  - Investigational Site Number 792202, Istanbul
  - Investigational Site Number 792204, Izmir
  - Investigational Site Number 792203, Izmir

REFERENCES:
- [Result] Derwahl KM, Bailey TS, Wernicke-Panten K, Ping L, Pierre S. Efficacy and Safety of Biosimilar SAR342434 Insulin Lispro in Adults with Type 2 Diabetes, Also Using Insulin Glargine: SORELLA 2 Study. Diabetes Technol Ther. 2018 Jan;20(1):49-58. doi: 10.1089/dia.2017.0281. Epub 2017 Dec 12. PMID 29232162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 103 centers in 12 countries. A total of 707 participants were screened between 14 January 2015 and 24 July 2015, of which 202 were screen failures. Screen failures were mainly due to glycated hemoglobin (HbA1c) level <6.5% or >10% at screening visit.
Pre-assignment Details: A total of 505 participants were randomized and treated in the study. Randomization was stratified by HbA1c at the screening visit (<8%, >=8%) and prior use of Humalog (Yes, No). Assignment to arms was done centrally using interactive voice/web response system in 1:1 ratio (SAR342434: Humalog).
Groups:
- SAR342434: SAR342434 100 U/mL SC injection before meals intake on top of QD Insulin Glargine, up to Week 26.
- Humalog: Humalog 100 U/mL SC injection before meals intake on top of QD Insulin Glargine, up to Week 26.
Period: Overall Study
Arm/Group | SAR342434 | Humalog
Started | 253 | 252
Completed | 228 | 230
Not Completed | 25 | 22
Not completed — Adverse Event | 7 | 7
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Other than specified above | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- SAR342434: SAR342434 100 U/mL subcutaneous (SC) injection before meals intake on top of once daily (QD) Insulin Glargine, up to Week 26.
- Total: Total of all reporting groups
Arm/Group | SAR342434 | Humalog | Total
Number analyzed (Participants) | 253 | 252 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.4) | 62.8 (8.9) | 62.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 120 | 237
  Male | 136 | 132 | 268
Previous meal time insulin [Count of Participants; unit: Participants]
  Humalog/Liprolog | 133 | 126 | 259
  NovoLog/NovoRapid | 119 | 124 | 243
  Both Humalog/Liprolog and NovoLog/NovoRapid | 1 | 1 | 2
  None of the above | 0 | 1 | 1
Randomization Strata of Screening HbA1c [Count of Participants; unit: Participants]
  <8 % | 105 | 104 | 209
  >=8 % | 148 | 148 | 296
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (4.8) | 32.1 (4.8) | 32.2 (4.8)
Duration of type 2 diabetes mellitus (T2DM) [Mean (Standard Deviation); unit: years] | 16.6 (7.93) | 17.52 (8.67) | 17.06 (8.31)
HbA1c % [Mean (Standard Deviation); unit: percentage of hemoglobin] | 8 (0.86) | 8.03 (0.91) | 8.01 (0.89)
Average Daily Basal Insulin Dose [Mean (Standard Deviation); unit: U/kg] — Population: Number of participants analyzed = participants with available data for specified measure.
  U/kg
    number analyzed (Participants) | 232 | 244 | 476
    (all) | 0.477 (0.265) | 0.458 (0.239) | 0.467 (0.252)
Average Daily Mealtime Insulin Dose [Mean (Standard Deviation); unit: U/kg] — Population: Number of participants analyzed = participants with available data for specified measure.
  U/kg
    number analyzed (Participants) | 231 | 243 | 474
    (all) | 0.449 (0.294) | 0.433 (0.315) | 0.441 (0.305)
Average Daily Total Insulin Dose [Mean (Standard Deviation); unit: U/kg] — Population: Number of participants analyzed = participants with available data for specified measure.
  U/kg
    number analyzed (Participants) | 230 | 242 | 472
    (all) | 0.927 (0.47) | 0.888 (0.449) | 0.907 (0.459)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Change in HbA1c was calculated by subtracting baseline value from Week 26 value. Adjusted least square means and standard errors were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data, using all post-baseline HbA1c data available during the 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on intent-to-treat (ITT) population that included all randomized participants, irrespective of compliance with the study protocol and procedures. Here, number of participants analyzed = participants with at least one post-baseline HbA1c assessment during the 6-month study period.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 239 | 246
percentage of HbA1c | -0.92 (0.051) | -0.85 (0.051)
Statistical Analysis 1: Comparison: SAR342434 vs Humalog; Analysis was performed using a MMRM approach with treatment groups, randomization strata, visit (Week 12, Week 26) and treatment-by-visit interaction as fixed categorical effects and baseline HbA1c value and baseline HbA1c value-by-visit interaction as continuous fixed covariates. An unstructured correlation matrix was used to model within-participant errors; Test type: Non-Inferiority — Non-inferiority of SAR342434 over Humalog was demonstrated if upper bound of 2-sided 95% confidence interval(CI) of difference between SAR342434 & Humalog was <0.3%.Inverse non-inferiority of Humalog over SAR342434 was tested using hierarchical step-down testing procedure: if non-inferiority of SAR342434 over Humalog was demonstrated,then inverse non-inferiority of Humalog over SAR342434 was tested and demonstrated if lower bound of 2-sided 95% CI of difference between SAR342434 & Humalog>-0.3%; Least Square (LS) Mean Difference = -0.07, 95% CI 2-sided [-0.215 to 0.067], Standard Error of Mean 0.072 — SAR342434 vs. Humalog

2. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and <=6.5% at Week 26
Description: Participants who had no available assessment for HbA1c at Week 26 were considered as non-responders.
Time Frame: Week 26
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 252
percentage of participants
  HbA1c <7.0% | 42.3 | 40.5
  HbA1c<=6.5% | 27.3 | 24.2

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: Change in FPG was calculated by subtracting baseline value from Week 26 value. Adjusted least squares means and standard errors were obtained from a MMRM approach to account for missing data, using all post-baseline FPG data available during the 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, number of participants analyzed = participants with at least one post-baseline FPG assessment during the 6-months study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 228 | 235
mmol/L | -0.62 (0.176) | -0.67 (0.176)

4. Secondary Outcome: Change in Mean 24-Hour Plasma Glucose Concentration From Baseline to Week 26
Description: The mean 24-hour plasma glucose concentration was calculated based on 7-point self-measured plasma glucose (SMPG) profiles with plasma glucose measurements before and 2-hours after each main meal and at bedtime. 7-point SMPGs were performed at least two times in a week before baseline, before visit Week 12 and before visit Week 26. Mean 24-hour plasma glucose concentration was calculated for each profile and then averaged across profiles performed in the week before a visit. Change in mean 24-hour plasma glucose concentration was calculated by subtracting baseline value from Week 26 value. Adjusted least squares means and standard errors were obtained from a MMRM to account for missing data, using all post-baseline data available during 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, number of participants analyzed = participants with at least one post-baseline mean 24-hour plasma glucose concentration assessment during 6-month study period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- SAR342434: SAR342434 100 U/mL SC injection before meals intake on top of QD Insulin Glargine up to Week 26.
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 201 | 210
mmol/L | -1 (0.137) | -0.91 (0.133)

5. Secondary Outcome: Change in Post Prandial Glucose (PPG) Excursion From Baseline to Week 26
Description: Plasma glucose excursions were calculated at breakfast, lunch and dinner for each 7-point SMPG profile, as 2-hour postprandial glucose (PPG) minus plasma glucose value obtained 30 minutes prior to start of the meal. Values of plasma glucose excursions at each visit were then calculated as average across the profiles performed in the week before the visit. Change in PPG excursions was calculated by subtracting baseline value from Week 26 value. Adjusted least squares means and standard errors were obtained from a MMRM to account for missing data, using all post-baseline data available during the 6-month period and adequate contrasts at Week 26.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, number analyzed in each row = participants with at least one post-baseline data during the 6-month period for specified categories.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 252
mmol/L
  At breakfast: number analyzed (Participants) | 194 | 204
  At breakfast | -0.72 (0.236) | -0.23 (0.228)
  At lunch: number analyzed (Participants) | 195 | 200
  At lunch | 0.06 (0.255) | 0.11 (0.25)
  At dinner: number analyzed (Participants) | 190 | 193
  At dinner | 0.11 (0.264) | -0.1 (0.264)

6. Secondary Outcome: Percentage of Participants With Hypoglycemia (Any Hypoglycemia, Documented Symptomatic Hypoglycemia and Severe Hypoglycemia)
Description: Percentage of participants with at least one treatment emergent hypoglycemia reported at any time of the day were reported. Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=70 mg/dL (3.9 mmol/L). Hypoglycemic episodes with plasma glucose of 54 mg/dL (<3.0 mmol/L) were also analyzed.
Time Frame: First dose of study drug up to 1 day after the last dose administration (maximum treatment exposure: 210 days)
Population: Analysis was performed on safety population that included all participants randomized and exposed to at least 1 dose of investigational medicinal product (IMP) (SAR342434 or Humalog), regardless of the amount of treatment administered.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 252
percentage of participants
  Any hypoglycemia | 68.4 | 74.6
  Severe hypoglycemia | 2.4 | 1.6
  Documented Symptomatic Hypoglycemia (<=3.9mmol/L) | 60.1 | 66.3
  Documented Symptomatic Hypoglycemia (<3.0mmol/L) | 28.9 | 27.4

7. Secondary Outcome: Percentage of Participants With Hypersensitivity Reactions and Injection Site Reactions
Description: Percentage of participants with hypersensitivity reactions and injection site reactions were reported.
Time Frame: First dose of study drug up to 1 day after the last dose administration (maximum treatment exposure: 210 days)
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 252
percentage of participants
  Any hypersensitivity reactions | 4 | 3.6
  Any injection site reactions | 0.4 | 1.6

8. Secondary Outcome: Percentage of Participants With Treatment-Emergent Anti-insulin Antibodies (AIAs)
Description: Participants with treatment-emergent AIA (incidence) were reported (as participants with treatment-boosted or treatment-induced AIAs). Participants with treatment-induced AIAs were participants who developed AIA following IMP administration (participants with at least one positive AIA sample at any time during on-treatment period, in those participants without pre-existing AIA or with missing baseline sample). Participants with treatment-boosted AIAs were participants with pre-existing AIAs that were boosted to a significant higher titer following IMP administration (participants with at least one AIA sample with at least a 4-fold increase in titers compared to baseline value at any time during on-treatment period, in those participants with pre-existing AIA).
Time Frame: First dose of study drug up to 1 day after the last dose administration (maximum treatment exposure: 210 days)
Population: Analysis was performed on anti-insulin antibody population that included all participants from the safety population with at least one AIA sample available for analysis during the 6-months on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 245 | 248
percentage of participants | 18.8 | 14.5

9. Other Pre Specified Outcome: Change in Daily Insulin Dose From Baseline to Week 26
Description: Change in daily insulin dose (basal, mealtime and total) was calculated by subtracting baseline value from Week 26 value.
Time Frame: Baseline, Week 26
Population: Analysis was performed on safety population. Here, number analyzed in each row = participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | SAR342434 | Humalog
Number analyzed (Participants) | 253 | 252
U/kg
  Basal insulin: number analyzed (Participants) | 196 | 218
  Basal insulin | 0.082 (0.133) | 0.071 (0.122)
  Mealtime insulin: number analyzed (Participants) | 197 | 218
  Mealtime insulin | 0.087 (0.209) | 0.08 (0.248)
  Total insulin: number analyzed (Participants) | 196 | 216
  Total insulin | 0.172 (0.296) | 0.151 (0.297)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Day 183) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment-emergent adverse events that is AEs that developed, worsened or became serious during the 'on treatment period' (time from first injection of IMP up to 1 day after the last injection of IMP).
Arm/Group | SAR342434 | Humalog
All-Cause Mortality (participants affected / at risk) | 1/253 | 2/252
Serious Adverse Events (participants affected / at risk) | 14/253 | 27/252
Other Adverse Events (participants affected / at risk) | 0/253 | 0/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAR342434 (N=253) | Humalog (N=252)
Angina pectoris (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Gliosis (Nervous system disorders) | 1 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.